CLINICAL TRIAL: NCT04660851
Title: Improving Diet Protein Intake in Middle-aged Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Responsible Party: Principal Investigator, Sareen Gropper, PhD, RDN, LDN, Professor, Florida Atlantic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1440147-1
Record Dates: First submitted 2020-10-16; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Dietary Habits
Keywords: Protein intake, coaching, strength
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coached (Experimental): 10 weeks of diet coaching
  Interventions: Behavioral: Coached
- Not-coached (No Intervention): No coaching provided

INTERVENTIONS:
Behavioral: Coached — 10-weeks of diet coaching weekly by telephone to improve dietary protein intake
  Arms: Coached

SUMMARY:
The study sought to examine the effectiveness of nutrition education with and without diet coaching on dietary protein intake and muscle mass, strength and function among a group of middle-aged women.

DETAILED DESCRIPTION:
The study sought to examine the effectiveness of nutrition education alone and with 10 weeks of diet coaching on dietary protein intake and muscle mass, strength and function among a group of middle-aged women.

ELIGIBILITY:
Inclusion Criteria:

* able to understand and respond to questions or instructions in English
* working telephone
* willingness to consume protein-containing animal products,
* willingness to make changes to the diet

Exclusion Criteria:

* self-reported information that they have been told by a medical doctor that they have kidney (renal) disease
* current or past history of a diagnosed eating disorder
* have an internal cardiac pacemaker/defibrillator or other metal-type implant present
* vegan dietary practices
* refusal to make changes to usual dietary protein intake
* usual dietary protein intake greater than 1.2 g per kg body weight

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Changes in dietary protein intake from baseline | 12 weeks
  Assessed changes in dietary protein intake from three 24-hour dietary recalls collected at baseline.

SECONDARY OUTCOMES:
Changes in muscle mass | 12 weeks
  Changes in muscle mass from baseline were measured using bioelectrical impedance analysis
Changes in upper body muscle strength | 12 weeks
  Changes in handgrip strength from baseline were measured using hand dynamometer
Changes in lower body muscle strength and function | 12 weeks
  Changes in 5-chair stand times from baseline were assessed
Changes in muscle function | 12 weeks
  Changes in 4 meter gait speed from baseline were assessed

CONTACTS AND LOCATIONS:
Overall Officials: Sareen S Gropper, PhD, Principal Investigator — Professor, College of Nursing, Florida Atlantic University
Locations (1):
- Florida Atlantic University, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No